CLINICAL TRIAL: NCT03304197
Title: How Does Altering the Composition of Ingested Fluids Affect Hydration Status Whilst Cycling?
Brief Title: Hydration and Exercise Performance in Cycling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 170614/A/01
Record Dates: First submitted 2017-09-13; First posted 2017-10-06 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Doubly-blinded & randomised using an online randomisation website.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dehydrated (Experimental): 90 minutes cycling, without the ingestion of any fluids, followed by a 15 minute cycling time trial test
  Interventions: Other: Dehydrated
- Hypotonic (Experimental): 90 minutes cycling, with the ingestion of six 250 ml carbohydrate (6g sucrose, 3g glucose) drinks, followed by a 15 minute cycling time trial test
  Interventions: Dietary Supplement: Hypotonic
- Isotonic (Experimental): 90 minutes cycling, with the ingestion of six 250 ml carbohydrate (6g glucose, 3g fructose) drinks, followed by a 15 minute cycling time trial test
  Interventions: Dietary Supplement: Isotonic
- Placebo (Experimental): 90 minutes cycling, with the ingestion of six 250 ml taste-matched water drinks, followed by a 15 minute cycling time trial test
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hypotonic — N/A: see arm description
  Arms: Hypotonic
Dietary Supplement: Isotonic — N/A: see arm description
  Arms: Isotonic
Dietary Supplement: Placebo — N/A: see arm description
  Arms: Placebo
Other: Dehydrated — N/A: see arm description
  Arms: Dehydrated

SUMMARY:
This study will evaluate the effects manipulating ingested fluids can have on hydration status and cycling performance. There will be 4 different conditions.

DETAILED DESCRIPTION:
Being dehydrated can decrease endurance exercise performance. The investigators wish to test which of three drinks is most effective at re-hydrating cyclists and if this affects performance. Subjects will undertake 4 tests: once dehydrated, once hydrated with water, once hydrated with a sports-specific drink, and once with an altered sports drink. Blood samples will be taken and expired gasses will be sampled at various time points throughout the tests for later analysis. A small amount of labelled water will be consumed with each drink, a technique which will allow us to quantify the absorption of each of the drinks.

ELIGIBILITY:
Inclusion Criteria:

* Highly trained cyclists (vo2max >55 ml/kg/min, PPO (peak power output) > 4 w/kg)
* Training at least 4 times a week
* Females must be taking an oral contraceptive, or using the contraceptive implant

Exclusion Criteria:

* Recent history of musculoskeletal injury
* Diagnosed cardiovascular disease
* Regular use of nutritional supplements that may interfere with the protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Absorption of fluid through the gut | To begin 10 minutes after the completion of the 90 minute steady-state cycle
  Absorption of drinks through the gut will be measured using 2 boluses of deuterated water. This will be consumed alongside 2 of the drinks, and blood samples will be used to quantify enrichment. Total body water calculations are required to provide corrections in equations related to D2O. H218O will be consumed in order to quantify total body water: this will be provided in a single bolus before each trial.

SECONDARY OUTCOMES:
Work done (kJ) during 15 minute cycling time-trial | Throughout the 90 minute steady-state cycle & the 15 minute time trial.
  Subjects will perform a cycle ergometer protocol that has been shown to be reproducible in athletes. Subjects will complete the time trial on a Lode Excalibur cycling ergometer. Software linked to this software will record work done and power output.

OTHER OUTCOMES:
Substrate utilisation | Throughout the 90 minute steady-state cycle
  Substrate utilisation will be calculated from data collected through a metabolic cart and its software. It will be measured during the 90-minute steady-state cycle for 4 periods of 3 minutes. Carbohydrate and lipid oxidation rates will be calculated using equations by Jeukendrup & Wallis (2005).
Plasma metabolites | Throughout the 90 minute steady-state cycle and time-trial
  A cannula will be used to draw blood from subjects at several time points. Whole blood samples will be analysed immediately for plasma glucose, plasma lactate, haemoglobin content, haematocrit and plasma volume. Remaining whole blood will be centrifuged immediately and its plasma split into aliquots and stored in a -20°C freezer. At the end of the trial, plasma samples will be moved to a -80°C freezer for later analysis for sodium, glycerol, and NEFA.
Heart rate | Throughout the 90 minute steady-state cycle and time-trial
  Heart rate will be measured throughout with the use of a heart rate monitor.
RPE (rating of perceived exertion) | Throughout the 90 minute steady-state cycle and time-trial
  RPE will be measured using the Borg Scale.
Core body temperature | Throughout the 90 minute steady-state cycle and time-trial
  Core temperature will be measured throughout with the use of an ingestible core-body temperature pill (HQ Inc, FL, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Davenport, MSc, Principal Investigator — The University of Exeter
Locations (1):
- School of Sports and Health Sciences, Exeter, Devon, United Kingdom